CLINICAL TRIAL: NCT06354296
Title: Comparison of the Accuracy of Different Intraocular Lens Power Calculation Formulas in Cataract Patients With Prior Radial Keratotomy
Status: Not yet recruiting | Type: Observational
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CAF2024
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Cataract
Keywords: cataract; RK surgery; formula
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Web-based Barret True K formula with no history formula has been proven to be a good choice for cataract patients after RK in several studies. The American society of cataract and refractive surgeons provides several IOL formulas for cataract patients who have undergone previous corneal refractive surgery. In cases where only IOL-Master data are available, Holladay 1 (Double-K) [Holladay 1 (D-K)] can be used for IOL power calculation in cataract patients with a history of RK. The traditional Haigis formula has also been shown to be effective for cataract patients after RK. To compare the accuracy of four intraocular lens (IOL) power calculation formulas in cataract patients after RK. They are Barrett True-K formula, Holladay 1(D-K) formula, Haigis formula, and MM formula.

DETAILED DESCRIPTION:
Myopia is the most common cause of distance vision impairment. The prevalence of myopia has increased dramatically in the past few decades, especially in China. Corneal refractive surgery is an effective method to correct adult myopia. Radial keratotomy (RK) is one of the corneal refractive surgeries developed in the 1980s. Thirty years ago, many myopic patients underwent RK. As patients age, more and more patients have cataracts requiring cataract extraction and intraocular lens (IOL) implantation. The selection of appropriate and accurate IOL is an important factor to improve patient satisfaction. Recent studies have compared the accuracy of the newly developed IOL formula in patients with previous RK cataract. However, as a country with myopia and myopia surgery, there is no similar study in China. In addition, most patients with cataract after RK had lost ocular data before RK surgery. For RK patients without previous ocular data, how to accurately calculate the IOL power is still a clinical challenge.

ELIGIBILITY:
Inclusion Criteria:

* Had a previous history of RK surgery
* IOL-Master is available
* There were no intraoperative and postoperative complications
* Obvious refraction was performed 1 to 6 months after cataract surgery

Exclusion Criteria:

* The investigator decided that it was not suitable for this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cataract after RK
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the IOL formula | Baseline
  To compare the accuracy of four intraocular lens (IOL) calculation formulas in cataract patients after radial keratotomy (RK). They are Barrett True-K formula, Holladay 1(D-K) formula, Haigis formula, and MM formula